CLINICAL TRIAL: NCT07206017
Title: Measuring Effects of High-fiber Dried Chicory Root on the Gut Microbiota of Patients With an Intermediate to High-risk Cutaneous Melanoma: an Explorative Study
Brief Title: Explorative Study on Addition of High-fiber Dried Chicory Root in Patients With an Intermediate to High-risk Cutaneous Melanoma.
Acronym: MELFIB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19789
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Melanoma, Stage II
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prebiotic dried chicory root (WholeFiber) (Experimental): Supplementing with WholeFiber for 6 weeks two times a day (10 g per portion). During 3 visits questionnaires, measurements and (blood and fecal) samples will be taken.
  Interventions: Other: prebiotic dried chicory root (WholeFiber)

INTERVENTIONS:
Other: prebiotic dried chicory root (WholeFiber) — Supplementing with WholeFiber for 6 weeks two times a day (10 g per portion).

SUMMARY:
Exploring the effect of supplementation with daily addition of prebiotic dried chicory root (WholeFiberTM) for 6 weeks on fecal SCFA levels, gut microbial composition and immune cell composition in minimal stage II A melanoma patients following surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* The participant understands the study and can provide written informed consent;
* The participant received surgical treatment of an intermediate to high-risk cutaneous melanoma (T2a/N1, T2b, T3a, T3b, T4a, T4b, N0 or N+, M0 stadium without evidence of disease);
* Being able to read and speak Dutch;
* Willing to come to the UMCG for practical reasons (visiting the study site);
* Willing to continue their regular lifestyle patterns during the study.

Exclusion Criteria:

* Receiving concurrent adjuvant treatment, adjuvant treatment after the study period is allowed.
* Having a medical history that may impact study outcomes, such as a diagnosis of diabetes mellitus type 2, heart disease, renal disease, autoimmune disease;
* Any clinically significant or unstable medical disorder involving the gut, including celiac disease, inflammatory bowel disease, short-bowel syndrome or acute/chronic pancreatitis;
* Having an ileostomy or colostomy, as this greatly impacts bowel function and gut microbial composition;
* Use of antibiotics in the 3 months prior participation in the study;
* Use of prednisolone or other immunosuppressive medication;
* Use of tube feeding or sib-feeding;
* Being pregnant or lactating;
* Participation in another interventional study at the same time;
* Unable or unwilling to comply to study rules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2027-09-14 (Estimated)

PRIMARY OUTCOMES:
Effect of a high fiber prebiotic vegetable (WholeFiber) on fecal SCFA levels | 6 weeks
  Effect of a high fiber prebiotic vegetable (WholeFiber) for 6 weeks on fecal SCFA levels in intermediate to high-risk cutaneous melanoma patients, with no concurrent adjuvant treatment. HPLC ion chromatography system (Metrohm AG, Herisau, Switzerland) will be used to determine the levels of SCFA. The concentrations of SCFA; butyrate, propionate, and acetate will be measured with a conductivity detector. SCFA will be measured at baseline, halfway intervention and after 6 weeks.

SECONDARY OUTCOMES:
Discovering the gut microbial composition changes | 6 weeks
  Discovering the gut microbial composition changes measured in intermediate to high-risk cutaneous melanoma patients with no concurrent adjuvant treatment, after using WholeFiber for 6 weeks. This analysis will be based on whole genome sequencing of fecal samples performed at the UMCG according to standardized protocol.
Exploring the effect of WholeFiber use | 6 weeks
  Exploring the effect of WholeFiber use for 6 weeks on immune functioning, stool patterns, fecal calprotectin levels and side effects in this patient group. Peripheral blood mononuclear cells (PBMCs) and bloodplasma will be isolated to determine immune cell composition before and after the intervention period. Fecal calprotectin will be determined using the respective ELISA kit (Thermo Fisher Scientific). Calprotectin is released when neutrophils enter the gut wall and are activated during the inflammatory process. Lastly, eating patterns, fiber intake before the interventional period, stool patterns and side effects will be identified using the Food Frequency Questionnaire, Bristol Stool Scale, Gastrointestinal Symptoms Rating Scale and Health Related Quality of Life questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: G. A.P. Hospers, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- UMCG, Groningen, Provincie Groningen, Netherlands

DOCUMENTS (2):
  • Study Protocol (2025-02-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT07206017/Prot_000.pdf
  • Informed Consent Form (2025-02-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT07206017/ICF_001.pdf